CLINICAL TRIAL: NCT01977391
Title: Association Between Mortality and Diabetes in Elderly Koreans: the South-West Seoul (SWS) Study
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Other Study IDs: SWS(mortality, DM)
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Apparently Healthy Elderly People; (Between 60-92 Years of Age)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Diabetes mellitus is known to increase the risk of premature death in the general population. In this study, the investigators examine the impact of body mass index (BMI) levels, waist circumference, and presence/absence of diabetes on all-cause and cardiovascular mortality in elderly Koreans.

DETAILED DESCRIPTION:
The investigators analyze follow-up data from the South-West Seoul (SWS) Study, a prospective observational cohort study of an elderly Korean population residing in Seoul, the metropolitan capital city of Korea.

Briefly, the study population was selected from four urban districts (Guro, Yangcheon, Gwanak and Gangseo) located in the south-west area of Seoul. A total of 1737 apparently healthy individuals (between 60 and 92 years of age) eventually participated in this survey starting in 1999. A follow-up examination was performed in 2002, and an additional 873 subjects who had not participated in the first examination were newly recruited.

After a median follow-up of 10 years, each subject's vital status or cause of death as of 31 December 2011 was determined after linking these cohort data with death certificate data from the Korean National Statistical Office. Terminology and codes from the International Classification of Disease, Tenth Revision (ICD-10), were used to classify the underlying cause of death due to cardiovascular disease (ICD-10 codes I00-I79), cancer (ICD-10 codes C00-C97) and others.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy individuals
* Over the age of 60 years

Exclusion Criteria:

* Those with a mismatched identification number
* Missing data regarding BMI, waist circumference, and presence of diabetes

Ages: 60 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects in South-West Seoul (SWS) study, a prospective observational cohort study of an elderly Korean population residing in Seoul, the metropolitan capital city of Korea.
Sampling Method: Probability Sample
Enrollment: 2263 (Actual)
Dates: Start 1999-08; Primary Completion 2002-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
All-cause and cardiovascular mortality in elderly Korean men and women according to BMI, waist circumference, and presence of diabetes | A median follow-up of 10 years

SECONDARY OUTCOMES:
Survival probability among study populations | A median follow-up of 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Univ. Guro Hospital, Seoul, South Korea

REFERENCES:
- [Background] Choi KM, Lee J, Kim DR, Kim SK, Shin DH, Kim NH, Park IB, Choi DS, Baik SH. Comparison of ADA and WHO criteria for the diagnosis of diabetes in elderly Koreans. Diabet Med. 2002 Oct;19(10):853-7. doi: 10.1046/j.1464-5491.2002.00783.x. PMID 12358874
- [Background] Choi KM, Lee J, Kim KB, Kim DR, Kim SK, Shin DH, Kim NH, Park IB, Choi DS, Baik SH; South-west Seoul Study. Factor analysis of the metabolic syndrome among elderly Koreans--the South-west Seoul Study. Diabet Med. 2003 Feb;20(2):99-104. doi: 10.1046/j.1464-5491.2003.00890.x. PMID 12581260
- [Background] Kim NH, Cho HJ, Kim YJ, Cho MJ, Choi HY, Eun CR, Kim JH, Yang SJ, Yoo HJ, Kim HY, Seo JA, Kim SG, Baik SH, Choi DS, Choi KM. Combined effect of high-normal blood pressure and low HDL cholesterol on mortality in an elderly Korean population: the South-West Seoul (SWS) study. Am J Hypertens. 2011 Aug;24(8):918-23. doi: 10.1038/ajh.2011.78. Epub 2011 Apr 28. PMID 21525969